CLINICAL TRIAL: NCT01379430
Title: Safety and Immunogenicity of Heterologous Prime-boost With the Candidate Malaria Vaccines AdCh63 ME-TRAP and MVA ME-TRAP in Healthy Adults in a Malaria Endemic Area
Brief Title: Safety and Immunogenicity of AdCh63 ME-TRAP and MVA ME-TRAP Vaccines in Malaria Endemic Areas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Kenya Medical Research Institute (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC040
Record Dates: First submitted 2011-06-10; First posted 2011-06-23 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Malaria
Keywords: Vaccine; Immune response
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Intramuscular arm
  Interventions: Biological: AdCh63 ME-TRAP followed by MVA ME-TRAP
- Group 2 (Experimental): Intradermal arm
  Interventions: Biological: AdCh63 ME-TRAP followed by MVA ME-TRAP

INTERVENTIONS:
Biological: AdCh63 ME-TRAP followed by MVA ME-TRAP — AdCh63 ME-TRAP 1x10^10 vp intramuscularly, MVA ME-TRAP 2x10^8 pfu intramuscularly
  Arms: Group 1
Biological: AdCh63 ME-TRAP followed by MVA ME-TRAP — AdCh63 ME-TRAP 5x10^10 vp intramuscularly, MVA ME-TRAP 2x10^8 pfu intradermal
  Arms: Group 2

SUMMARY:
The purpose of this trial is to assess the safety and immunogenicity of AdCh63 ME-TRAP and MVA ME-TRAP candidate vaccines in healthy adult volunteers in a malaria endemic region. The regime proposed in this trial has protected non-immune volunteers against sporozoite challenge in clinical trials performed by Oxford, and so may be protective against naturally acquired infection in Kenya.The study population will comprise 30 healthy adult males aged 18-50.

The investigators do not propose to include a placebo group. At this stage the investigators objective is to describe the safety profile in a small number of individuals, and the confidence intervals for the proportion of individuals with a particular event would be too wide for meaningful comparison with a placebo group. Immunogenicity will be judged by comparison with baseline.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult males aged 18-50 years in good health.
* Will remain resident in the study area for the study duration

Exclusion Criteria:

* Clinically significant history of the following conditions; skin disorder (eczema, etc.), allergy, symptomatic immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness.
* History of splenectomy
* Haemoglobin less than 9.0 g/dl
* Clinically significant abnormalities of laboratory screening tests (full blood count, ALT, creatinine levels, urine dipstick examination for blood and protein).
* Blood transfusion within one month of the beginning of the study
* History of vaccination with previous experimental malaria vaccines
* Administration of any other vaccine or immunoglobulin within two weeks before vaccination.
* Current participation in another clinical trial, or within 12 weeks of this study
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial.
* Likelihood of travel away from the study area
* HIV positive.
* History of contact dermatitis (due to the use of a potentially irritant disinfectant that may be present in trace amounts in the AdCh63 ME-TRAP vaccine, see the investigators brochure for details, attached)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity of AdCh63 ME-TRAP followed by MVA ME-TRAP in adults in Kenya. | Participants will be followed for the duration of the study, an expected average of 12 months
  To assess safety and reactogenicity of AdCh63 ME-TRAP followed by MVA ME-TRAP in adults in Kenya by recording local and systemic solicited and unsolicited adverse events

SECONDARY OUTCOMES:
Immunogenicity of vaccines | Participants will be followed for the duration of the study, an expected average of 12 months
  To evaluate the immunogenicity of AdCh63 ME-TRAP followed by MVA ME-TRAP in adults in Kenya by assessing induced antibody and T cell response to the vaccine insert.
Immunogenicity of Vaccines | Participants will be followed for the duration of the study, an expected average of 12 months
  To compare the use of intra-muscular and intra-dermal MVA ME-TRAP

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI/Wellcome Trust Programme, Centre for Geographic Medicine Research - Coast, Kilifi, Kenya

REFERENCES:
- [Derived] Ogwang C, Afolabi M, Kimani D, Jagne YJ, Sheehy SH, Bliss CM, Duncan CJ, Collins KA, Garcia Knight MA, Kimani E, Anagnostou NA, Berrie E, Moyle S, Gilbert SC, Spencer AJ, Soipei P, Mueller J, Okebe J, Colloca S, Cortese R, Viebig NK, Roberts R, Gantlett K, Lawrie AM, Nicosia A, Imoukhuede EB, Bejon P, Urban BC, Flanagan KL, Ewer KJ, Chilengi R, Hill AV, Bojang K. Safety and immunogenicity of heterologous prime-boost immunisation with Plasmodium falciparum malaria candidate vaccines, ChAd63 ME-TRAP and MVA ME-TRAP, in healthy Gambian and Kenyan adults. PLoS One. 2013;8(3):e57726. doi: 10.1371/journal.pone.0057726. Epub 2013 Mar 19. PMID 23526949